CLINICAL TRIAL: NCT02472119
Title: Wheat Flour Subjected to Microbial Transglutaminase Enzymatic Treatment in the Presence of Lysine Ethyl Ester for Alimentary Use in the Treatment of Celiac Disease.
Brief Title: Wheat Flour Treatment With Microbial Transglutaminase and Lysine Ethyl Ester: New Frontiers in Celiac Disease Treatment.
Acronym: WHETMIT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Antonio Picarelli, Medical Doctor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 672/10 Rif. 1907 / 22.07.2010
Record Dates: First submitted 2015-06-03; First posted 2015-06-15 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-06

CONDITIONS: Celiac Disease
Keywords: Celiac disease; Gluten-free diet; Wheat flour treatment; Microbial transglutaminase; Lysine Ethyl Ester; Celiac Disease Treatment
MeSH Terms: conditions — Celiac Disease | interventions — Diet, Gluten-Free

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- rusks made with treated flour (Experimental): Gluten-free diet adding rusks (100g / day) produced with commercial wheat flour enzymatically treated with mTGasi and lysine ethyl ester.
  Interventions: Dietary Supplement: rusks made of wheat flour enzymatically treated; Dietary Supplement: Gluten-free diet
- rusks made with not-treated flour (Active Comparator): Gluten-free diet adding rusks (100g / day) produced with untreated wheat flour.
  Interventions: Dietary Supplement: rusks made of wheat flour not enzimatically modified; Dietary Supplement: Gluten-free diet

INTERVENTIONS:
Dietary Supplement: rusks made of wheat flour enzymatically treated — 100 g of rusks obtained from commercial wheat flour enzymatically treated with mTGasi and lysine ethyl ester, every day for 3 months
  Arms: rusks made with treated flour
Dietary Supplement: rusks made of wheat flour not enzimatically modified — 100 g of rusks obtained from commercial wheat flour NOT enzymatically treated with mTGasi and lysine ethyl ester, every day for 3 months
  Arms: rusks made with not-treated flour
Dietary Supplement: Gluten-free diet — gluten-free diet

SUMMARY:
Celiac disease is one of the most common forms of food intolerance (prevalence 1/200). The disease occurs in genetically predisposed individuals after ingestion of foods containing gluten. Celiac patients can suffer from severe malabsorption syndrome, mainly characterized by diarrhea and weight loss. The only therapeutic approach currently recognized is a life-long gluten-free diet.

Specific regions of gluten molecule become recognizable by lymphocytes and activate them, due to changes made by tissue transglutaminase. These changes consist in the conversion of specific residues of glutamine into glutamic acid. The consequence is an increased binding affinity between gluten and histocompatibility molecule (HLA-DQ2), localized on the surface of the "antigen presenting cells" (APC); the exposure of the fragments of modified gluten on the surface of APC is a phenomenon that eventually activates T lymphocytes.

Recent studies on modified gluten confirmed the hypothesis that it is possible to block the presentation of gluten to lymphocytes by means of lysine ethyl ester binding exclusively to those gluten regions responsible for lymphocyte activation.

The enzymatic treatment is performed directly on flour instead of extracted gluten, maintaining the same anti-inflammatory effectiveness.

The procedure uses a food-grade enzyme, the microbial transglutaminase (mTGasi) isolated from Streptoverticillium mobarensis, able to catalyze the formation of intermolecular "cross-links" that modify the functional properties of the products.

Objective of the study is to validate the ability of the enzyme treatment of wheat flour with mTGasi and lysine ethyl ester to block the toxic effect of gluten in celiac patients.

DETAILED DESCRIPTION:
Celiac disease is one of the most common forms of food intolerance (prevalence 1/200). The disease occurs in genetically predisposed individuals after ingestion of foods containing wheat gluten and similar proteins found in other common cereals such as barley and rye. Celiac patients can suffer from severe malabsorption syndrome, mainly characterized by diarrhea, weight loss and growth retardation. The only therapeutic approach currently recognized is a life-long gluten-free diet.

Specific regions of gluten molecule become recognizable by lymphocytes and activate them, due to changes made by tissue transglutaminase. These changes consist in the conversion of specific residues of glutamine (Q) into glutamic acid (E). The consequence is an increased binding affinity between gluten and histocompatibility molecule (HLA-DQ2), localized on the surface of the "antigen presenting cells" (APC); the exposure of the fragments of modified gluten on the surface of APC is a phenomenon that eventually activates T lymphocytes.

Recent studies on modified gluten confirmed the hypothesis that it is possible to block the presentation of gluten to lymphocytes by means of lysine ethyl ester binding exclusively to those gluten regions responsible for lymphocyte activation.

Specifically, it is possible to perform the enzymatic treatment directly on flour instead of extracted gluten, maintaining the same anti-inflammatory effectiveness. The final procedure consists in dissolving the flour in water in the presence of appropriate concentrations of enzyme and lysine ethyl ester, maintaining the suspension in constant motion for two hours at room temperature.

The procedure uses a food-grade enzyme, the microbial transglutaminase (mTGasi) isolated from Streptoverticillium mobarensis, already used for the preparation of food. The mTgasi is able to catalyze the formation of intermolecular "cross-links" modifying the functional properties of the products through the aggregation and polymerization of proteins. The peculiar method identified by our laboratory reduces the possibility of cross-links between proteins: consequently, minimal changes involve the gluten structure and, consequently, the visco-elastic properties of the dough.

Objective of the study is to validate the ability of the enzyme treatment of wheat flour with mTGasi and lysine ethyl ester to block the toxic effect of gluten in celiac patients.

ELIGIBILITY:
Inclusion Criteria:

INCLUSION CRITERIA

* diagnosis of celiac disease according to ESPGHAN criteria: class III according to Marsh-Oberhuber classification, clear response to gluten-free diet, serological antiendomysium and antitransglutaminase antibodies positive results before GFD;
* HLA DQ2-DQ8 positive results;
* gluten-free diet from at least one year;
* negative serology from at least 1 year;

EXCLUSION CRITERIA

* inflammatory bowel diseases;
* tumors;
* infectious liver disease;
* renal impairment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-06; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in IgA anti-tissue transglutaminase (anti-tTG) antibodies at 30 days | After 1 month
  Proof of any positivization of specific serological antibodies for celiac disease. Results quantified by an ELISA reader at 450 nm (A450nm) is expressed in U/mL and the antibody level 10 U/mL was used as a cutoff value to identify anti-tTG positive results.
Change from baseline in IgA anti-tissue transglutaminase (anti-tTG) antibodies at 60 days | After 2 months
  Proof of any positivization of specific serological antibodies for celiac disease. Results quantified by an ELISA reader at 450 nm (A450nm) is expressed in U/mL and the antibody level 10 U/mL was used as a cutoff value to identify anti-tTG positive results.
Change from baseline in IgA anti-tissue transglutaminase (anti-tTG) antibodies at 90 days | After 3 months
  Proof of any positivization of specific serological antibodies for celiac disease. Results quantified by an ELISA reader at 450 nm (A450nm) is expressed in U/mL and the antibody level 10 U/mL was used as a cutoff value to identify anti-tTG positive results.
Change from baseline in IgA anti-endomysium antibodies (EMA) at 30 days | After 1 month
  Test used to confirm serological activation of celiac disease. IgA EMA were searched in sera diluted 1:5 by indirect immunofluorescence analysis on cryostat sections of monkey esophagus. The results are expressed as ''positive/negative''.
Change from baseline in IgA anti-endomysium antibodies (EMA) at 60 days | After 2 months
  Test used to confirm serological activation of celiac disease. IgA EMA were searched in sera diluted 1:5 by indirect immunofluorescence analysis on cryostat sections of monkey esophagus. The results are expressed as ''positive/negative''.
Change from baseline in IgA anti-endomysium antibodies (EMA) at 90 days | After 3 months
  Test used to confirm serological activation of celiac disease. IgA EMA were searched in sera diluted 1:5 by indirect immunofluorescence analysis on cryostat sections of monkey esophagus. The results are expressed as ''positive/negative''.
Pathologic variations in histologic analysis from baseline | After 3 months, or in case of serum anti-tTG IgA/EMA IgA positive results
  Proof of duodenal mucosa histological alterations induced by celiac disease, consisting in altered (<3:1) villous height/crypt depth ratio and increased (>25) intraepithelial lymphocytes per 100 intestinal epithelial cells, according to Marsh-Oberhuber classification.

SECONDARY OUTCOMES:
Presence of bloating at baseline | At baseline
  Evaluation of bloating intensity is reported according to the Visual Analog or Analogue Scale (VAS), with a range of 0-10.
Presence of abdominal pain at baseline | At baseline
  Evaluation of abdominal pain intensity is reported according to the Visual Analog or Analogue Scale (VAS), with a range of 0-10.
Presence of diarrhea at baseline | At baseline
  Evaluation of diarrhea intensity is reported according to the Visual Analog or Analogue Scale (VAS), with a range of 0-10.
Presence of asthenia at baseline | At baseline
  Evaluation of asthenia intensity is reported according to the Visual Analog or Analogue Scale (VAS), with a range of 0-10.
Variation of bloating from baseline at 30 days | After 1 month
  Evaluation of bloating intensity is reported according to the Visual Analog or Analogue Scale (VAS), with a range of 0-10.
Variation of abdominal pain from baseline at 30 days | After 1 month
  Evaluation of abdominal pain intensity is reported according to the Visual Analog or Analogue Scale (VAS), with a range of 0-10.
Variation of diarrhea from baseline at 30 days | After 1 month
  Evaluation of diarrhea intensity is reported according to the Visual Analog or Analogue Scale (VAS), with a range of 0-10.
Variation of asthenia from baseline at 30 days | After 1 month
  Evaluation of asthenia intensity is reported according to the Visual Analog or Analogue Scale (VAS), with a range of 0-10.
Variation of bloating from baseline at 60 days | After 2 months
  Evaluation of bloating intensity is reported according to the Visual Analog or Analogue Scale (VAS), with a range of 0-10.
Variation of abdominal pain from baseline at 60 days | After 2 months
  Evaluation of abdominal pain intensity is reported according to the Visual Analog or Analogue Scale (VAS), with a range of 0-10.
Variation of diarrhea from baseline at 60 days | After 2 months
  Evaluation of diarrhea intensity is reported according to the Visual Analog or Analogue Scale (VAS), with a range of 0-10.
Variation of asthenia from baseline at 60 days | After 2 months
  Evaluation of asthenia intensity is reported according to the Visual Analog or Analogue Scale (VAS), with a range of 0-10.
Variation of bloating from baseline at 90 days | After 3 months
  Evaluation of bloating intensity is reported according to the Visual Analog or Analogue Scale (VAS), with a range of 0-10.
Variation of abdominal pain from baseline at 90 days | After 3 months
  Evaluation of abdominal pain intensity is reported according to the Visual Analog or Analogue Scale (VAS), with a range of 0-10.
Variation of diarrhea from baseline at 90 days | After 3 months
  Evaluation of diarrhea intensity is reported according to the Visual Analog or Analogue Scale (VAS), with a range of 0-10.
Variation of asthenia from baseline at 90 days | After 3 months
  Evaluation of asthenia intensity is reported according to the Visual Analog or Analogue Scale (VAS), with a range of 0-10.

CONTACTS AND LOCATIONS:
Locations (1):
- Sapienza University - Policlinico Umberto I, Rome, Italy, Italy

REFERENCES:
- [Background] Branski D, Fasano A, Troncone R. Latest developments in the pathogenesis and treatment of celiac disease. J Pediatr. 2006 Sep;149(3):295-300. doi: 10.1016/j.jpeds.2006.06.003. No abstract available. PMID 16939736
- [Background] Nilsen EM, Jahnsen FL, Lundin KE, Johansen FE, Fausa O, Sollid LM, Jahnsen J, Scott H, Brandtzaeg P. Gluten induces an intestinal cytokine response strongly dominated by interferon gamma in patients with celiac disease. Gastroenterology. 1998 Sep;115(3):551-63. doi: 10.1016/s0016-5085(98)70134-9. PMID 9721152
- [Background] Molberg O, Mcadam SN, Korner R, Quarsten H, Kristiansen C, Madsen L, Fugger L, Scott H, Noren O, Roepstorff P, Lundin KE, Sjostrom H, Sollid LM. Tissue transglutaminase selectively modifies gliadin peptides that are recognized by gut-derived T cells in celiac disease. Nat Med. 1998 Jun;4(6):713-7. doi: 10.1038/nm0698-713. PMID 9623982
- [Background] Gianfrani C, Siciliano RA, Facchiano AM, Camarca A, Mazzeo MF, Costantini S, Salvati VM, Maurano F, Mazzarella G, Iaquinto G, Bergamo P, Rossi M. Transamidation of wheat flour inhibits the response to gliadin of intestinal T cells in celiac disease. Gastroenterology. 2007 Sep;133(3):780-9. doi: 10.1053/j.gastro.2007.06.023. Epub 2007 Jun 20. PMID 17678925
- [Background] Yokoyama K, Nio N, Kikuchi Y. Properties and applications of microbial transglutaminase. Appl Microbiol Biotechnol. 2004 May;64(4):447-54. doi: 10.1007/s00253-003-1539-5. Epub 2004 Jan 22. PMID 14740191
- [Background] Fink ML, Chung SI, Folk JE. gamma-Glutamylamine cyclotransferase: specificity toward epsilon-(L-gamma-glutamyl)-L-lysine and related compounds. Proc Natl Acad Sci U S A. 1980 Aug;77(8):4564-8. doi: 10.1073/pnas.77.8.4564. PMID 6107907
- [Background] Catassi C, Fabiani E, Iacono G, D'Agate C, Francavilla R, Biagi F, Volta U, Accomando S, Picarelli A, De Vitis I, Pianelli G, Gesuita R, Carle F, Mandolesi A, Bearzi I, Fasano A. A prospective, double-blind, placebo-controlled trial to establish a safe gluten threshold for patients with celiac disease. Am J Clin Nutr. 2007 Jan;85(1):160-6. doi: 10.1093/ajcn/85.1.160. PMID 17209192
- [Background] Picarelli A, Di Tola M, Sabbatella L, Anania MC, Calabro A, Renzi D, Bai JC, Sugai E, Carroccio A, Di Prima L, Bardella MT, Barisani D, Ribes-Koninckx C, Aliaga ED, Gasparin M, Bravi E; Multicentre Organ Culture System Study Group. Usefulness of the organ culture system in the in vitro diagnosis of coeliac disease: a multicentre study. Scand J Gastroenterol. 2006 Feb;41(2):186-90. doi: 10.1080/00365520510024151. PMID 16509042
- [Background] Picarelli A, Maiuri L, Frate A, Greco M, Auricchio S, Londei M. Production of antiendomysial antibodies after in-vitro gliadin challenge of small intestine biopsy samples from patients with coeliac disease. Lancet. 1996 Oct 19;348(9034):1065-7. doi: 10.1016/S0140-6736(96)03060-7. PMID 8874458
- [Derived] Marino M, Casale R, Borghini R, Di Nardi S, Donato G, Angeloni A, Moscaritolo S, Grasso L, Mazzarella G, Di Tola M, Rossi M, Picarelli A. The effects of modified versus unmodified wheat gluten administration in patients with celiac disease. Int Immunopharmacol. 2017 Jun;47:1-8. doi: 10.1016/j.intimp.2017.03.012. Epub 2017 Mar 23. PMID 28343108